CLINICAL TRIAL: NCT03230461
Title: Can Rescuers Accurately Deliver Subtle Changes to Chest Compression Depth if Recommended by Future Guidelines?
Brief Title: Estimation of CPR Chest Compression Depth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 19575
Record Dates: First submitted 2017-07-21; First posted 2017-07-26 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Arrest
Keywords: CPR; Basic life support
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Prospective, randomised.
Who Masked: Participant, Investigator
Masking Description: Participants and researchers are blinded to the actual depth achieved during each CPR run.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Target compression depth 4.0-5.0 cm (Experimental): The rescuer is asked to perform two minutes of chest compressions on a manikin, aiming to compress to the target depth at a rate of 100-120/min
  Interventions: Behavioral: Compression depth
- Target compression depth 4.5-5.5 cm (Experimental): The rescuer is asked to perform two minutes of chest compressions on a manikin, aiming to compress to the target depth at a rate of 100-120/min
  Interventions: Behavioral: Compression depth
- Target compression depth 5.0-6.0 cm (Experimental): The rescuer is asked to perform two minutes of chest compressions on a manikin, aiming to compress to the target depth at a rate of 100-120/min
  Interventions: Behavioral: Compression depth

INTERVENTIONS:
Behavioral: Compression depth

SUMMARY:
Optimal chest compression depth during CPR is 4.56cm which is at variance with the current guidelines of 5.0-6.0cm. A change in guidelines is only worthwhile if healthcare professionals can accurately judge a subtle reduction in chest compression depth during CPR by a relatively small amount.

DETAILED DESCRIPTION:
Chest compression depth and rate during cardiopulmonary resuscitation (CPR) are important predictors of return of spontaneous circulation and survival following cardiac arrest. Stiell et al (2014) found optimal survival at a compression depth of 4.56cm, which is at variance with the current guidelines of 5.0-6.0cm. A change in guidelines is only likely to improve survival rates if healthcare professionals can accurately implement these subtle depth modifications into the basic life support (BLS) algorithm. This study aims to determine if healthcare professionals can accurately judge compression depth without real-time feedback.

ELIGIBILITY:
Inclusion Criteria:

* NHS professionals (staff or students), who have successfully completed a hospital-accredited basic life support (BLS) course, including a practical CPR component.

Exclusion Criteria:

* Pregnancy, significant medical illness or injury that would impair delivery of chest compressions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Compression to target window depth | Two minutes
  Mean compression depth

SECONDARY OUTCOMES:
Compression to target rate | Two minutes
  Mean compression rate

CONTACTS AND LOCATIONS:
Overall Officials: Charles Deakin, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Available on request